CLINICAL TRIAL: NCT06023875
Title: An Open, Single-center, Phase II Trial of Cadonilimab Combined With Platinum-containing Dual-agent Neoadjuvant Therapy for Locally Advanced Operable Head and Neck Squamous Cell Carcinoma
Brief Title: Neoadjuvant Cadonilimab in Combination With Cisplatin and Nab-paclitaxel in Resectable Head and Neck Squamous Cell Carcinoma
Acronym: NCCCNRHNSCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuekui Liu (Other)
Responsible Party: Sponsor-Investigator, Xuekui Liu, chief physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-FXY-011-HNC
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Locally Advanced Operable
Keywords: head and neck squamous cell carcinoma; Cadonilimab; neoadjuvant therapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Patients with locally advanced operable head and neck squamous cell carcinoma
  Interventions: Drug: Cadonilimab; Drug: Docetaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Cadonilimab — Cadonilimab 10mg/kg. The drug was administered every 3 weeks (Q3W), and 21 days (Q3W) was a treatment cycle. The treatment regimen is recommended for three cycles until the researchers determine that the subjects cannot continue to benefit, until the disease progression (PD), the toxicity cannot be tolerated, the treatment is delayed by more than 14 days, or the patient withdraws the informed consent form or dies.
  Other Names: AK104
Drug: Docetaxel — Docetaxel 75mg/m2. Intravenous infusion was given every 3 weeks (Q3W), and 21 days (Q3W) was a treatment cycle. Treatment regimen is recommended for 3 cycles.
Drug: Cisplatin — Cisplatin 60mg/m2. Intravenous infusion was given every 3 weeks (Q3W), and 21 days (Q3W) was a treatment cycle. Treatment regimen is recommended for 3 cycles.

SUMMARY:
This study is a single arm phase ll trial including 30 patients with T2N2-3M0、T3-4N0-3M0 (lll-V) head and neck squamous cell carcinoma (HNSCC) eligible forresection, who receive neo-adjvuant Cadonilimab combined with cisplatin and Nab.paclitaxel.This proposed study will evaluate the efficacy and safety of preoperativeadministration of Cadonilimab combined with chemotherapy in Head and Neck Squamous Cell Carcinoma (HNSCC) who are about to undergo surgery.

DETAILED DESCRIPTION:
In this study, eligible subject will be enrolled into study arm to accept study treatment objective response rate will be the primary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed primary head and neck squamous cell carcinoma confirmed by histology and/or cytology (excluding diagnostic therapy).
2. Clinical stage: T2N2-3M0, T3-4N0-3M0 (III-IV) (AJCC 8th edition staging).
3. Age: 18 to 70 years.
4. PS score (see Appendix Table 1; performance status score of 0 or 1).
5. Patients evaluated by a head and neck oncologist as resectable with no distant metastases.
6. Patients with at least one measurable lesion according to RECIST version 1.1 criteria.
7. Patients' toxicities assessed according to CTCAE version 4.03 criteria.
8. Patients with normal organ function (heart, brain, lungs, kidneys) and suitable for surgery:

   1. Hematology: White blood cells ≥ 4000/μL, neutrophils ≥ 2,000/μL, hemoglobin ≥ 9 g/dL, platelets ≥ 100,000/μL;
   2. Liver function: Bilirubin ≤ 1.5 times the upper limit of normal (ULN) (patients with known Gilbert's disease and serum bilirubin levels ≤ 3 times ULN can be included), AST and ALT ≤ 3 times ULN, alkaline phosphatase ≤ 3 times ULN; albumin ≥ 3 g/dL;
   3. Renal function: Serum creatinine ≤ 1.5 times ULN or creatinine clearance ≥ 60 mL/min according to Cockcroft-Gault formula.
9. Consent to provide archived tumor tissue samples or undergo biopsy for collection of tumor lesion tissue (at least 3 unstained FFPE pathological slides, if deemed insufficient for PD-L1 IHC testing by the central laboratory, an additional 3 unstained FFPE pathological slides should be provided) to be sent to the central laboratory for PD-L1 immunohistochemistry (IHC) testing (preferably using recently obtained tumor tissue samples). Tumor lesions planned for biopsy should not be used for assessing target lesions of the disease unless no other suitable lesions for biopsy are available. Patients have signed an informed consent form, are willing and able to comply with the study's visit, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. History of severe hypersensitivity reactions to components of other monoclonal antibodies, CTLA4, or PD-1 antibodies.
2. Patients with known or suspected autoimmune diseases, including dementia and epileptic seizures.
3. Recurrence, distant metastasis, or the inability to undergo surgery as assessed by a head and neck physician.
4. Abnormal coagulation function: (PT > 16s, APTT > 53s, TT > 21s, Fib < 1.5g/L), bleeding tendency, or currently on anticoagulant or thrombolytic therapy.
5. Severe heart disease, pulmonary dysfunction, patients with heart or lung function below Grade 3 (including Grade 3).
6. Laboratory values not meeting relevant criteria within 7 days prior to enrollment.
7. Previous use of anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-PD-L2 antibodies, or anti-CTLA-4 antibodies (or any other antibodies targeting T cell co-stimulation or checkpoint pathways).
8. Pre-existing conditions requiring long-term use of immunosuppressive drugs or a need for systemic or local use of corticosteroids at immunosuppressive doses prior to enrollment.
9. HIV-positive individuals; HBsAg-positive individuals with positive HBV DNA copy number (quantitative test ≥ 1000 cps/ml); positive chronic hepatitis C blood screening (HCV antibody positive).
10. Traditional herbal medicine used for anti-tumor purposes within 4 weeks before randomization.
11. Active or prior history of documented inflammatory bowel disease (such as Crohn's disease, ulcerative colitis, or chronic diarrhea).
12. Women of childbearing potential with a positive pregnancy test and breastfeeding women.
13. Known active pulmonary tuberculosis (TB). Subjects suspected of having active TB need clinical evaluation for exclusion.
14. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
15. Severe infection occurring within 4 weeks before the first administration, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia.
16. Subjects planning major surgery within 30 days after the first dose of AK104 in combination with platinum-containing dual-agent therapy (as determined by the investigator), or not yet fully recovered from prior surgery. Local surgical procedures (such as placement of a systemic port and prostate biopsy) are allowed provided that the surgery is completed at least 24 hours before the first dose of the study treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 9 weeks
  overall response rate

SECONDARY OUTCOMES:
PCR | 9 weeks
  Pathological Complete Response
MPR | 9 weeks
  Major Pathological Response
DCR | 2 years
  Disease Control Rate
PFS | 2 years
  progression-free survival
OS | 5 years
  Overall survival
Adverse Events Graded By Ctcae V5.0 | 90 days after the first dose of study treatment
  Percentage of adverse events that are possibly, probably or definitely related to study treatment per Criteria for Adverse Events version 5 (CTCAE v5.0).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, 651 Dongfeng East Road, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, 651 Dongfeng East Road, Guangzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao F, Li Y, Fang Q, Lin R, Zhao Z, Xu P, Yan H, Zhang X, Jiang K, Zhou J, Chen C, Lu L, Han F, Li Z, Wu D, Liu X. Cadonilimab (a PD-1/CTLA-4 Bispecific Antibody) plus Neoadjuvant Chemotherapy in Locally Advanced Head and Neck Squamous Cell Carcinoma: A Phase II Clinical Trial. Clin Cancer Res. 2025 Sep 15;31(18):3876-3885. doi: 10.1158/1078-0432.CCR-25-1445. PMID 40705040